CLINICAL TRIAL: NCT02418793
Title: A Phase 1/2a, Open-Label, Multicenter, Dose Escalation Study to Assess the Safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) Profile of a Long Acting Recombinant FVIIa (MOD-5014) in Adult Men With Hemophilia A or B
Brief Title: A Study of a Long-Acting r-Factor 7a (Factor VIIa) in Adult Men With Hemophilia A or B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-5-001
Record Dates: First submitted 2015-03-31; First posted 2015-04-16 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Hemophilia; Factor VII; Factor VIIa; Inhibitors; Long Acting
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Dose Cohort 1 (Experimental): Lowest MOD-5014 dose tested in the study
  Interventions: Drug: MOD-5014
- Dose Cohort 2 (Experimental): MOD-5014 Dose cohort 2
  Interventions: Drug: MOD-5014
- Dose Cohort 3 (Experimental): MOD-5014 Dose cohort 3
  Interventions: Drug: MOD-5014
- Dose Cohort 4 (Experimental): MOD-5014 Dose cohort 4
  Interventions: Drug: MOD-5014
- Dose Cohort 5 (Experimental): MOD-5014 Dose cohort 5
  Interventions: Drug: MOD-5014
- Dose Cohort 6 (Experimental): Highest MOD-5014 dose tested in the study
  Interventions: Drug: MOD-5014

INTERVENTIONS:
Drug: MOD-5014 — Long Acting Factor VIIa

SUMMARY:
The purpose of the current Phase 1/2a single dose, dose-escalating study is to evaluate the acute safety, pharmacokinetics (PK) and pharmacodynamics (PD) properties of MOD-5014 in adult subjects with moderate/severe congenital hemophilia A or B. This will be a single-dose, open label, dose-escalating study. Each dose cohort will be concluded by a safety review, following which escalation to the next dose cohort will be approved.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate or severe congenital Hemophilia A or B with or without inhibitors

Exclusion Criteria:

* Diagnosis of any coagulation disorder other than Hemophilia A or B
* Receipt of any immunomodulatory therapy within 3 months prior to screening, with the exception of Hepatitis C or HIV therapy
* Have had, within one month prior to study drug administration, a major surgical procedure (e.g. orthopedic, abdominal) or have an elective surgery planned within the study period
* Use of any anticoagulant for arterial/venous obstructions and/or atrial fibrillation within 7 days prior to first study drug administration
* Malignancy within past 5 years (excluding non-melanoma skin cancer)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Composite safety and tolerability parameters as measured by adverse events, electrocardiograms (ECG), laboratory results, vital signs and injection site reactions | 30 days
  To assess the acute safety and tolerability of single intravenous (IV) administration of escalating MOD-5014 doses in hemophilic subjects with and without inhibitors.

SECONDARY OUTCOMES:
Pharmacokinetic Profile | 14 days
  To evaluate the pharmacokinetic profile (MOD-5014 serum levels; Area Under the Curve (AUC); Cmax; Tmax; T1/2) of single IV administration of escalating MOD-5014 doses in hemophilic subjects with and without inhibitors.

OTHER OUTCOMES:
Pharmacodynamic Profile (evaluate the pharmacodynamic response (FVIIa clotting activity, coagulation parameters) of single IV administration of escalating MOD-5014 doses) | 14 days
  To evaluate the pharmacodynamic response (FVIIa clotting activity, coagulation parameters) of single IV administration of escalating MOD-5014 doses in hemophilic subjects with and without inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Ben-Bashat, Study Director — OPKO Health, Inc.
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Rush University Medical Center, Chicago, Illinois
  - Bleeding & Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Presbyterian Shadyside, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - The Gulf States Hemophilia and Thrombophilia Center, Houston, Texas